CLINICAL TRIAL: NCT07139093
Title: Testing of an Interface for Synchronizing tACS-DBS With a Phase-locked-loop
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: University of Twente (Other); University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PV7207_1; SCHW 2023/2-1 (Other Grant/Funding Number: German Research Foundation)
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Deep Brain Stimulation; Parkinson's Disease (PD)
Keywords: deep brain stimulation; transcranial alternating current stimulation; EEG; synchronization; brain-computer interface

STUDY DESIGN:
Intervention Model Description: Active DBS and active tACS with different phase-lags (at least 4: 0°, 90°, 180°, 270°)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- phase-lags (Experimental): Device: phase-lags
  * DBS will be applied at a fixed frequency between 15-30 Hz in one hemisphere only using the contact(s) of the clinical DBS settings. The amplitude of the electrode in the other hemisphere will be set to 0mA.
  * tACS will be applied closed-loop at the same frequency as DBS; with 4 phase lags relative to the DBS pulse (0°, 90°, 180°, 270°). tACS will be administered using the neuroConn DC-STIMULATOR PLUS.
  * EEG will be measured during this intervention with an analog (Digitimer) amplifier.
  Interventions: Device: DBS-coupled tACS

INTERVENTIONS:
Device: DBS-coupled tACS — tACS will be applied in a phase-coupled manner, so that tACS and DBS are synchronized

SUMMARY:
The investigators aim to test an interface to phase-lock transcranial alternating current stimulation (tACS) and deep brain stimulation (DBS) for future studies investigating the effects of different time-lags between DBS and tACS on the behavioural and neural level. To test if the interface works in patients with DBS, the investigators record EEG during synchronized tACS-DBS in several patients. The investigators hypothesize that they can apply tACS at the desired phase-lags relative to DBS pulses and confirm this with EEG measurements of the DBS and tACS artifact.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent by the patient
* Age 35 - 85
* patient groups: Parkinson's disease, essential tremor, dystonia
* >3 months after surgery for DBS

Exclusion Criteria:

* Epilepsy or history of seizures
* Existence of heart pacemaker or other metal implants in the body (except DBS)
* Pregnancy

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Phase-locking success | during stimulation procedure
  The investigators will measure the temporal precision of the locking of the tACS to the DBS pulses should be seen. To this end, the tACS-DBS artifact and the triggers given from the interface device will be analysed offline in MATLAB.

CONTACTS AND LOCATIONS:
Overall Officials: Bettina C. Schwab, PhD, Principal Investigator — UKE Hamburg
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided